CLINICAL TRIAL: NCT00624845
Title: Double-Blind, Multicenter, Study Comparing the Efficacy and Safety of OMS103HP
Brief Title: Double-Blind, Multicenter, Study Comparing the Efficacy and Safety of OMS103HP With Vehicle Irrigation Solution in Subjects Undergoing Meniscectomy
Acronym: C07-004
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Omeros Corporation (Industry)
Responsible Party: Gregory Demopulos, MD, CEO,CMO, Omeros Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C07-004
Record Dates: First submitted 2008-02-19; First posted 2008-02-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Postoperative Pain
Keywords: Meniscectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — OMS 103HP

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug (Experimental)
  Interventions: Drug: OMS103HP
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: OMS103HP — Maximum 6 bags of OMS103HP irrigation solution
  Arms: Drug
Drug: Vehicle — Maximum of 6 bags of vehicle irrigation solution
  Arms: Vehicle

SUMMARY:
The purpose of this study is to assess the benefit of OMS103HP for Injection (OMS103HP) compared with vehicle irrigation solution for prevention of pain and pain relief in subjects undergoing meniscectomy. The pain relief is assessed based on Visual Analog Scale (VAS) Pain Scores in the immediate 24-hour postoperative period and for seven days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has voluntarily signed informed consent form, including HIPAA Authorization.
2. Subject is ≥ 18 and ≤ 75 years of age.
3. Subject is in good general health with a traumatic or degenerative meniscal cartilage injury (full tear) that occurred at least 14 days prior to the day of arthroscopic surgery.
4. Subject is undergoing unilateral meniscectomy.
5. Subject's physical examination is within normal limits or examination is clinically nonsignificant as determined by the Investigator, and subject is in good general health.
6. Subject's laboratory evaluations are within normal limits or evaluations are clinically nonsignificant as determined by the Investigator.
7. Subject, if female and of childbearing potential (i.e., not surgically sterilized or post-menopausal greater than one year) agrees to use an effective method of birth control for the duration of her study involvement.
8. Subject is at minimal risk from anesthesia and is classified according to the American Society of Anesthesiologists Physical Status Classification as either PS-1 (a normal healthy patient) or PS-2 (a patient with mild systemic disease that results in no functional limitation). See Appendix VI.
9. Subject agrees to refrain from taking the excluded medications listed in Exclusion Criteria through postoperative Day 7 (except for authorized analgesic medications) unless written permission has been granted by Omeros.
10. Subject is able to be proficient in the use of the ePRO device (documented at the site).

Exclusion Criteria:

1. Subject with significant arthritis (>2 on the Kellgren-Lawrence Scale).
2. Subject with a history of reactive synovial disease.
3. Subject with current, or history of, complex regional pain syndrome (Type I, i.e., reflex sympathetic dystrophy, or Type II, i.e., causalgia), chronic pain, attendance at a chronic pain clinic, or neurologic disorder associated with any sensory deficit of the lower extremities.
4. Subject with current, or history of fibromyalgia.
5. Subject taking ANY ANALGESIC (including salicylates, opioids, propoxyphene, etc.) on the day of surgery from 12:00 A.M. until after the procedure, except for medications authorized by the Investigator or delegated staff.
6. Subject taking any of the following medications within the stated time frames prior to the day of surgery.

   1. Amitriptyline within 30 days
   2. More than two doses of sumatriptan, (or any other drug in the triptan class), ondansetron, or other prescription serotonergic or histaminic drug within 14 days
   3. More than two doses of any oral, parenteral, or intravenous steroids (e.g., dexamethasone for antiemetic prophylaxis) within 3 months
   4. More than two doses of oxymetazoline or other nasal decongestant/cold/cough/allergy medication (including loratadine) within 7 days
   5. More than two doses of ketoprofen or other NSAID (including COX-2 inhibitors) within 7 days (except for piroxicam, as indicated below)
   6. Subject who has taken more than two doses of opioid pain medication within the prior seven days of surgery or chronic use of opioid pain medications for greater than 6 weeks within the prior year
   7. More than two doses of piroxicam within 14 days
   8. Subject with a history of intra-articular corticosteroid injection in the operative knee within the two months prior to the meniscectomy
7. Subject expected to undergo any of the following procedures concurrent with meniscectomy:

   1. Arthroscopic patellar tendon debridement
   2. Patellar alignment
   3. Lateral or retinacular release
   4. Excision synovectomy (minor synovectomy to improve arthroscopic visualization is acceptable)
   5. Concurrent ligamentous procedure
   6. Microfracture
   7. Abrasion arthroplasty
   8. Chondral transplantation
   9. Use of more than three portals
8. Subject with allergies to any of the individual ingredients in OMS103HP, to related compounds (e.g., other NSAIDs or tricyclic antidepressants), or to opioid analgesics.
9. Subject who is pregnant or breast-feeding.
10. Subject with Worker's Compensation claim(s) under dispute or mediation.
11. Subject with history of drug or alcohol abuse.
12. Subject who has taken or used an investigational drug or device within 30 days prior to the day of surgery.
13. Subject with a history or presence of systemic disease (renal, hepatic, psychiatric, etc.), which in the opinion of the Medical Monitor and the Principal Investigator, may place the subject's health at risk by participation in the study.
14. Subject who is expected to receive a regional block for analgesia for this procedure.
15. Subject who is considered by the Investigator for any reason to be an unsuitable candidate for receipt of an investigational drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the mean VAS at 24 hours postoperatively. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Scott Houston, Study Director — Omeros Corporation
Locations (8):
- United States (8):
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - Visions Clinical Research, Tucson, Arizona
  - Kerlan-Jobe Orthopaedic Clinic - Westchester, Los Angeles, California
  - Advanced Orthopedic and Sports Medicine Specialists, Aurora, Colorado
  - Colorado Orthopedic Consultants, Englewood, Colorado
  - Greater Chesapeake Orthopaedic Associates, Baltimore, Maryland
  - University Orthopedics Center, State College, Pennsylvania
  - Unlimited Research, San Antonio, Texas